CLINICAL TRIAL: NCT05780021
Title: Evaluation of the Effectiveness of a MOTIVational Support Program After Multidisciplinary Functional Rehabilitation in Chronic Low Back Pain
Brief Title: Motivational Support Program in Chronic Low Back Pain After Multidisciplinary Functional Rehabilitation
Acronym: EMOTIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210077; 2022-A00828-35 (Other: ANSM)
Record Dates: First submitted 2023-01-23; First posted 2023-03-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Multidisciplinary function rehabilitation; Motivational Support Program Emotiv

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention): The patients will have the usual care
- Motivational Support Program Emotiv (Experimental): The patients will have the motivational support program
  Interventions: Behavioral: Motivational Support Program Emotiv

INTERVENTIONS:
Behavioral: Motivational Support Program Emotiv — A motivational support program including a motivational and self-assessment remote application in the form of a Smartphone application for chronic low back pain patients after multidisciplinary functional rehabilitation.
  Arms: Motivational Support Program Emotiv

SUMMARY:
Chronic low back pain (CLBP) is a major public health problem. Multidisciplinary functional rehabilitation program (FRP), which give patients the skills to better manage pain and return to physical activity, are effective in the short term. In the medium and long term, due to lack of motivation, two thirds of patients stop their physical activity again, causing them to fall back into the vicious circle of pain. Investigators hypothesise that a remote assessment and motivational support program (MSP) based on an application, piloted by a care coordinator, could allow the continued improvement of symptoms and activities observed after the FRP programs, and thus limit the consequences of CLBP for the patient and society. The main objective of this study is to evaluate the effect of the motivational support program EMOTIV, on disability and pain at one year, in chronic low back pain patients who have benefited from a FRP program.

DETAILED DESCRIPTION:
Multidisciplinary functional rehabilitation program (FRP) have shown their efficacy in disabilitie patient suffering from Chronic low back pain (CLBP). Unfortunately, at medium and long term two thirds of patients stop their physical activity due to lack of motivation. These patients then fall back into their painful vicious circle. Investigators hypothesis that motivational support program (MSP) based on an application, piloted by a care coordinator could increase the motivation to continue physical activity and thus limit the consequences of CLBP for the patient and society. The main objective is to evaluate the impact of a MSP (EMOTIV) on pain and functional abilities assessed according to the COMI scale (Core Outcome Measure Index), 12 months after a FRP in patients with LPBC. This program is compared to usual care as currently done. The secondary criteria concern: physical, neuropsychological and medico-economical criteria. This is a multicentre, cluster randomized trial. All adult patient suffering from low back pain, having finished a FRP and possessing a smartphone, will be included. Investigators plan to include 150 patients in 6 centres. The duration of the inclusion period is 12 months; The duration of participation of each subject is 24 months. Inclusion will be on the last day of the FRP program. The Follow-up in consultation is scheduled at 3, 12 and 24 months with evaluation of usual criteria (physical, self-questionnaires, and advice on the practice of physical activities depending on what is achieved). In Pitie salpetriere center only, patients will have in addition: lumbar MRI at 3 and 12 months; central pain awareness assessment. The activity of patients in the MSP group will be recorded continuously par EMOTIV App; pain, mental health and days off every week and self-questionnaires at 1, 2 and 6 months. The primary analysis of all endpoints will be performed in the intent-to-treat population, i.e. all patients randomized to the study. The COMI score will be compared between the 2 randomized groups by a linear mixed model.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* Disabling chronic low back pain: chronic painful patient, that is to say suffering from pain for more than 3 months, having interrupted all physical activity because of low back pain and have an indication for a FRP for low back pain.
* Having reached the end of an FRP program
* Possession of a smartphone
* Fluency in French (writing, reading)
* Health insurance coverage (beneficiary or beneficiary) except State Medical Aid.
* Patient Informed Consent Signature

Exclusion Criteria:

* Pregnant woman
* Patient refusal
* Patient deprived of liberty and patient under legal protection measure (guardianship, guardianship)
* Patient participating to another interventional search

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Difference in disability and pain between the experimental (SHP) and control (usual care) groups, measured with the Core Outcome Measure Index (COMI) scale at 12 months. | 12 months after completion of the multidisciplinary functional rehabilitation program
  The Core Outcome Measure Index (COMI) was developed from requirements of international back pain experts. According to European experts, the COMI should currently be recommended in assessment of chronic low back pain. This questionnaire assesses pain and disability in low back pain. It includes 9 items and its score is between 0 and 10. Higher scores is the worse outcome.

SECONDARY OUTCOMES:
Evolution of pain | At 3 months, 12 months and 24 months
  Pain will be measured by a Visual Analogic Scale (VAS) with a question about lumbar pain over the last 7 days. Minimum and maximum values are 0 and 100.
Evolution of flexibility | At 3 months, 12 months and 24 months
  Flexibility will be evaluated by measuring the hand-to-ground distance
Evolution of muscular endurance | At 3 months, 12 months and 24 months
  Muscular endurance will be assessed by measuring Shirado (abdominal endurance). Its score is between 0 and no limit. 0 is the worse outcome.
Evolution of muscular endurance | At 3 months, 12 months and 24 months
  Muscular endurance will be assessed by measuring Sorensen (spinal extensor endurance). Its score is between 0 and no limit. 0 is the worse outcome.
Evolution of disability and pain | At 3 months, 12 months and 24 months
  Disability and pain will be assessed by the Core Outcome Measure Index (COMI) questionnaire. Its score is between 0 and 10. Higher scores is the worse outcome.
Evolution of endurance and sports performance (VO2 max) | At 3 months, 12 months and 24 months
  Endurance and sports performance will be assessed on the treadmill
Evolution of the intensity of physical activity | At 3 months, 12 months and 24 months
  Intensity of physical activity will be assessed by the IPAQ (International Physical Activity Questionnaire). Scoring a high level of physical activity on the IPAQ means the physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
Evolution of muscular trophicity in the 2 groups | At 3 months and 12 months
  Muscular trophicity will be done by the measurement of the cross-sectional area (CSA) of the extensor muscles at the level of the upper and lower plateaus of L4 at the lumbar spine
Evolution of the level of anxiety and depression | At 3 months, 12 months and 24 months
  Level of anxiety and depression will be assessed by the HAD (Hospital Anxiety and Depression) scale.
  14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores (maximum and worse of each score equal 21)
Evolution of the level of central pain awareness | At inclusion, 3 months, 12 months and 24 months
  Two parameters will be used, in accordance with international recommendations on Quantitative Sensory Testings : the pain pressure threshold using an algometer, at a distance from the painful area (forearm), and the temporal summation by repeating a painful stimulus with a calibrated needle (PinPrick)
Medico-economic analysis | At 3 months, 12 months and 24 months
  The elements for the medico-economic analysis will be collected on the basis of a questionnaire validated in French. The data collected are : - consultations in general medicine and rheumatology as part of the usual follow-up of patients, - biological or imaging examinations carried out for the spinal problem, - medicinal treatments (drugs, infiltrative procedures) and non-medicinal treatments (physiotherapy, others) carried out for the spinal problem, - any hospitalizations related to the spinal problem
Cost of care (i.e, health resource use and related costs or direct costs) | At 3 months, 12 months and 24 months
  Health resource use will be quantified by the number of consultations, biologic and imaging workups, hospitalisations with their motives, and the list of treatments taken by the patients. It will be valued on the basis of the tariffs of the National Health Insurance Fund (CNAM). Health resource use related costs will be expressed in Euros
Cost of care (i.e, health resource use and related costs or direct costs) | At 3 months, 12 months and 24 months
  Health resource use will be quantified by the number of consultations, biologic and imaging workups, hospitalisations with their motives, and the list of treatments taken by the patients. It will be valued using data from the Common Classification of Medical Acts (CCAM). Health resource use related costs will be expressed in Euros
Cost of care (i.e, health resource use and related costs or direct costs) | At 3 months, 12 months and 24 months
  Health resource use will be quantified by the number of consultations, biologic and imaging workups, hospitalisations with their motives, and the list of treatments taken by the patients. It will be valued using data from the Nomenclature of Medical Biology Acts (NABM). Health resource use related costs will be expressed in Euros
Cost of care (i.e, health resource use and related costs or direct costs) | At 3 months, 12 months and 24 months
  Health resource use will be quantified by the number of consultations, biologic and imaging workups, hospitalisations with their motives, and the list of treatments taken by the patients. It will be valued using data from the national scale of costs (ENC) for hospitalisations. Health resource use related costs will be expressed in Euros
Sick leave days | At 3 months, 12 months and 24 months
  The number of working days off work will be elicited
Productivity loss (i.e, sick leave-related costs or indirect costs) | At 3 months, 12 months and 24 months
  Sick leave days will be valued on the basis of the average daily salaries published each year by the French National Institute of Statistics (INSEE, www.insee.fr). It will be expressed in Euros.
Satisfaction with the program | At 3 months, 12 months and 24 months
  Satisfaction with the program will be measured by a Visual Analogic Scale (VAS). Minimum and maximum values are 0 and 100. The better score is 100.
Adherence to the program | At 3 months, 12 months and 24 months
  Adherence to the program will be evaluated on the number of connection (minimum value 0 and no maximum)
Adherence to the program | At 3 months, 12 months and 24 months
  Adherence to the program will be evaluated on the time of connection (minimum value 0 and no maximum)
Adherence to the program | At 3 months, 12 months and 24 months
  Adherence to the program will be evaluated on number of reminders necessary by the coordinator in case of non connection and/or non attendance at the follow-up (minimum value 0 and non maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Violaine FOLTZ, Dr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.